CLINICAL TRIAL: NCT04005911
Title: Evaluation of Non-Contact Respiratory Rate Monitor in Post-Surgical Subjects
Brief Title: Non-Contact Respiratory Rate Monitoring
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Robert Thiele, MD, Associate Professor, University of Virginia
Other Study IDs: 21353
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Hypoxia
Keywords: Post-surgical
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-Surgical: Patients who underwent surgery and were admitted to the PACU
  Interventions: Device: Themography

INTERVENTIONS:
Device: Themography — Using a FLIR camera, a thermographic recording will be taken of the patient while breathing. Simultaneously, the research investigator will record the thoracic impedance-based respiratory rate as well as manually count respirations in one minute.

SUMMARY:
The purpose of this study is to compare thermographic estimates of respiratory rate to manual counting (visual inspection) and thoracic impedance-based methods. Thermographic methods rely on detection of temperature changes in the nose and mouth that occur as room temperature air passes through the nose and mouth during ventilation, and may offer a non-invasive means of measuring respiratory rate without requiring any patient contact.

ELIGIBILITY:
Inclusion Criteria:

* Underwent surgery at the University of Virginia
* Able to provide verbal consent to participate in the study

Exclusion Criteria:

* Unable to provide verbal consent to participate in the study
* Youth
* Prisoners

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Post-surgical patients in the PACU at the University of Virginia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-18 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Agreement between manually calculated respiratory rate and thermographic respiratory rate | 5 minutes
  Agreement between manually calculated respiratory rate and thermographic respiratory rate using the Limits of Agreement approach

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided